CLINICAL TRIAL: NCT00301847
Title: A Phase 2 Study of Sorafenib (BAY 43-9006) in Metastatic Renal Cell Cancer to the Brain
Brief Title: Sorafenib in Treating Patients With Kidney Cancer That Has Spread to the Brain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02689; UCCRC-14227; NCI-7296; CDR0000462558 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2006-04

CONDITIONS: Kidney Cancer; Metastatic Cancer
Keywords: tumors metastatic to brain; recurrent renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Neoplasm Metastasis; Brain Neoplasms; Carcinoma, Renal Cell | interventions — Sorafenib

ARMS (1):
- Arm I (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate

INTERVENTIONS:
Drug: sorafenib tosylate

SUMMARY:
This phase II trial is studying how well sorafenib works in treating patients with kidney cancer that has spread to the brain. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the partial and minor response rate in patients with renal cell carcinoma (RCC) metastatic to the brain treated with sorafenib.

SECONDARY OBJECTIVES:

I. Determine the toxicity of sorafenib in patients with RCC metastatic to the brain.

II. Determine whether the effect of sorafenib on RCC metastatic to the brain is similar to its effect on non-brain metastatic sites.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed renal cell carcinoma metastatic to the brain
* Measurable disease in the brain
* Meets 1 of the following criteria:

  * No prior brain-specific therapy AND no CNS symptoms referable to the brain lesion(s) (with or without concurrent steroid therapy)
  * CNS symptoms referable to the brain lesion(s) AND received primary therapy for the brain lesion(s)

PATIENT CHARACTERISTICS:

* Blood pressure < 140/90 mm Hg on 2 separate occasions, taken at least 24 hours apart, within the past 6 weeks (patients on stable anti-hypertensive regimens allowed)
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Bilirubin < 1.5 times upper limit of normal (ULN)
* ALT/AST < 2.5 times ULN
* Estimated glomerular filtration rate > 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow pills or comply with an oral treatment regimen
* No history of a bleeding diathesis or requirement for full-dose anticoagulation
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib
* No clinical or radiologic evidence of bowel obstruction or perforation
* No other uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* More than 4 weeks since prior radiotherapy to sites outside of the brain and recovered
* More than 8 weeks since prior standard external-beam radiotherapy to the brain unless there is evidence of in-brain progression
* No prior complete surgical resection or radiosurgery of all known brain metastases unless there is evidence of in-brain progression
* No prior sorafenib, sunitinib malate, bevacizumab, or any other agent targeting the platelet-derived growth factor receptor (PDGFR) or vascular endothelial growth factor receptor (VEGFR) kinase cascade
* No other concurrent investigational agents
* No concurrent enzyme-inducing anti-seizure medications, including phenytoin, phenobarbital, carbamazepine, or primidone

  * Concurrent non-enzyme-inducing anti-seizure medications allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent hematopoietic growth factors except erythropoietin
* No concurrent ketoconazole, itraconazole, or ritonavir
* No concurrent grapefruit juice
* No concurrent Hypericum perforatum (St. John's wort)
* No concurrent chemotherapy
* No concurrent hormonal therapy except steroids for adrenal failure and/or control of CNS edema or hormones for non-disease related conditions (e.g., insulin for diabetes)
* No concurrent palliative radiotherapy
* No other concurrent anticancer therapy
* Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Response rate by RECIST radiologic measurements every 8 weeks

SECONDARY OUTCOMES:
Safety by Common Toxicity Criteria version 3.0 every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Walter M. Stadler, MD, FACP, Principal Investigator — University of Chicago
Locations (12):
- United States (12):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin